CLINICAL TRIAL: NCT03245424
Title: Expanded Access Program for Ivosidenib (AG-120) Monotherapy in Patients With Relapsed or Refractory Acute Myeloid Leukemia With an IDH1 Mutation
Brief Title: Ivosidenib Expanded Access Program in Relapsed/Refractory AML With an IDH1 Mutation
Status: Approved for marketing | Type: Expanded Access
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AG120-C-010
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Acute Myeloid Leukemia; Relapsed Adult AML; Relapsed Pediatric AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ivosidenib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: ivosidenib (AG-120) — Patients will receive ivosidenib 500 mg by mouth once daily on 28-day cycles

SUMMARY:
To provide access to ivosidenib monotherapy to patients with relapsed or refractory acute myeloid leukemia (AML) with an isocitrate dehydrogenase 1 (IDH1) mutation.

DETAILED DESCRIPTION:
Study Conduct:

Patients who are eligible for enrollment will be entered into the study. Patients will receive ivosidenib 500 mg by mouth once daily on 28-day cycles until disease progression, unacceptable toxicity, physician or subject decision to discontinue, the subject proceeds to hematopoietic stem cell transplant, the subject dies, or until the study closes. Patients who achieve complete remission, undergo stem cell transplant, and then relapse can come back onto the study after consultation with the Medical Monitor. Enrollment into the study will close should ivosidenib be granted marketing authorization. If the study terminates for other reasons, access to drug will be assessed based on the rationale for termination.

Clinical Assessments:

All patients will have baseline assessments performed to confirm eligibility. Thereafter, treatment and assessments will be per routine standard of care at the investigational site and documentation will be maintained at the study site in the patient chart. Should study drug be discontinued, it is recommended that the patient return at least 28 days after receiving the last dose of study drug for a safety evaluation.

Safety assessments should be performed at intervals per institutional standard of care for patients taking ivosidenib. These assessments should include, but are not limited to: pregnancy tests, ECG, clinical lab assessments, vital signs and physical exam findings, and assessment of adverse events of special interest (AESIs)/serious adverse events (SAEs). Toxicity severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥12 years of age and weigh at least approximately 100 lbs.
2. Have AML with relapsed or refractory disease.
3. Have documented IDH1 R132 gene-mutated disease. (IDH1 mutation status will be based on local evaluation.)
4. Be able to understand and willing to sign an informed assent/consent. A legally authorized representative may consent on behalf of a patient who is otherwise unable to provide informed consent, if acceptable to and approved by the site and/or site's Institutional Review Board (IRB).
5. Have Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 3.
6. Have platelet count ≥20,000/µL. (Transfusions to achieve this level are allowed.) Patients with a baseline platelet count of <20,000/µL due to underlying malignancy are eligible with Medical Monitor approval.
7. Have adequate hepatic function as evidenced by:

   * Serum total bilirubin ≤1.5 × upper limit of normal (ULN), unless considered due to Gilbert's disease or leukemic involvement;
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤3.0 × ULN, unless considered due to leukemic involvement.
8. Have adequate renal function as evidenced by:

   • Creatinine clearance >30 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR) estimation: (140 -Age) x (weight in kg) x (0.85 if female)/72 x serum creatinine
9. Be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy, or other therapy intended for the treatment of cancer.
10. Female patients with reproductive potential must agree to undergo medically supervised pregnancy tests prior to starting study drug. The first pregnancy test will be performed at screening (within 7 days prior to first study drug administration); the second will be performed on the day of the first study drug administration and must be confirmed negative prior to dosing. Patients with reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy or tubal occlusion or who have not been naturally postmenopausal (i.e., who have not menstruated at all) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). Females of reproductive potential, as well as fertile men and their partners who are female of reproductive potential, must agree to use two effective forms of contraception (including at least one barrier form) from the time of giving informed assent/consent, during the study, and for 90 days (both females and males) following the last dose of AG-120. Effective forms of contraception are defined as hormonal oral contraceptives, injectables, patches, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal ligation, condoms with spermicide, or male partner sterilization.

Exclusion Criteria:

1. Are eligible to participate in a clinical trial or for whom potentially curative anticancer therapy is available.
2. Have previously received prior treatment with a mutant-specific IDH1 inhibitor and progressed on therapy.
3. Have undergone HSCT within 60 days of the first dose of ivosidenib, or patients on immunosuppressive therapy post HSCT at the time of screening, or with clinically significant graft-versus-host disease (GVHD). (The use of a stable dose of oral steroids post HSCT and/or topical steroids for ongoing skin GVHD is permitted with Medical Monitor approval.)
4. Have received systemic anticancer therapy or radiotherapy <14 days prior to their first day of study drug administration. (Hydroxyurea is allowed prior to enrollment and after the start of ivosidenib for the control of peripheral leukemic blasts in patients with leukocytosis [white blood cell {WBC}] counts >30,000/μL.)
5. Have received an investigational agent <14 days prior to their first day of study drug administration. In addition, the first dose of ivosidenib should not occur before a period ≥5 half-lives of the investigational agent has elapsed.
6. Are taking known strong CYP3A4 inducers or sensitive CYP3A4 substrate medications with a narrow therapeutic window, unless they can be transferred to other medications within ≥ 5 half-lives prior to dosing or unless the medications can be properly monitored during the study.
7. Are taking P-glycoprotein (P-gp) transporter-sensitive substrate medications with a narrow therapeutic window, unless they can be transferred to other medications within ≥5 half-lives prior to dosing or unless medications can be properly monitored during the study.
8. Are pregnant or breast feeding.
9. Have an active severe infection that requires anti-infective therapy or with an unexplained fever >38.5°C during Screening visits or on their first day of study drug administration (at the discretion of the Investigator, patients with tumor fever may be enrolled).
10. Have known hypersensitivity to any of the components of ivosidenib.
11. Have had New York Heart Association Class III or IV congestive heart failure (Appendix 14.2), myocardial infarction, unstable angina, and/or stroke.
12. Have a heart-rate corrected QT interval using Fridericia's method (QTcF) ≥ 470 msec or any other factor that increases the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome). Patients with prolonged QTcF interval in the setting of bundle branch block may participate in the study.
13. Have active hepatitis B or C. Patients with human immunodeficiency virus (HIV) infection are allowed provided their disease is under control on anti-retroviral therapy and that precautions are taken to modify their HAART regimen to minimize ivosidenib drug interactions. Such subjects should be monitored for a change in dosage requirements for the concomitant HAART drug when co-administering ivosidenib.
14. Have any other medical or psychological condition, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed assent/consent, cooperate, or participate in the study.
15. Have immediately life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult